CLINICAL TRIAL: NCT03310814
Title: Building New Nutrigenomics Technology Interface Tools for Consumers and Health Professionals
Brief Title: An Intervention to Develop Interface Tools for Nutrigenomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kwantlen Polytechnic University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Karen Davison, Principal Investigator, Kwantlen Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 500692 - 16
Record Dates: First submitted 2017-08-29; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Adult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized nutrition intervention (Experimental): Participant receives gene-test results plus personalized nutrition information from a registered dietician
  Interventions: Other: Personalized nutrition
- Usual nutrigenomics intervention (Placebo Comparator): Participant receives usual nutrigenomics intervention (direct-to-consumer)
  Interventions: Other: Personalized nutrition

INTERVENTIONS:
Other: Personalized nutrition — Receives individualized nutrition information

SUMMARY:
This study compares the efficacy of a non-practitioner assisted direct-to-consumer (DTC) self-driven approach to nutrigenomics versus a personalized practitioner-led method. The secondary aims are to use this data combined with participant feedback to generate more effective nutrigenomics-based products.

DETAILED DESCRIPTION:
While nutrition is a widely accepted tool for the prevention of long-term health conditions, current approaches have not adequately reduced chronic disease morbidity. Nutrigenomics has great potential, however, it is complicated to implement. There is a need for products, derived from nutrigenomics, which are easily understood, accessible and utilized. The primary objective of this study is to compare the efficacy of a non-practitioner assisted direct-to-consumer (DTC) self-driven approach to nutrigenomics versus a personalized practitioner-led method. The secondary aims are to use this data combined with participant feedback to generate more effective nutrigenomics-based products.

Methods:

This 4-month study used a mixed-methods design that included: 1) a phase 1 randomized control trial that examined the effectiveness of a multi-faceted, nutrition-based gene test (components assessed included the major nutrients, food tolerances, food taste and preferences, and vitamins) in changing health behaviours; followed by 2) qualitative investigation that explored participants' experiences. The study recruited 57 healthy males and females (35-55 years) randomized as a 2:1 ratio where 38 received the intervention (gene-test results plus personalized nutrition report) and 19 were assigned to the control group (gene-test results report emailed). Both groups received follow-up emails with nutrition-related tips and reminders. The primary outcomes of interest measures included changes in diet (nutrients, healthy eating index), self-efficacy, quality of life and anthropometrics (BMI, waist:hip) measured at baseline, post-intervention (3 and 6 weeks), and the final visit. After the study has been completed, participants in the control group will also receive their personalized nutrition report.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 35-55 years.
2. Ability to understand sign an informed consent and to give a buccal DNA swab.
3. Willing to improve their health.
4. Medically stable. Subjects diagnosed with diet-related chronic disease were able to enroll in the study, provided that their condition was stabilized or well controlled for at least six months at the time of the baseline visit. Determination of stabilized medical condition was based on established clinical guidelines (e.g., Canadian Diabetes Association Clinical Guidelines and Canadian Cardiovascular Society Guidelines).

Exclusion Criteria:

1. Currently on a therapeutic or restrictive diet (e.g., Atkins).
2. Diagnosis of 2 or more chronic diseases or unstable chronic disease as deemed by accepted clinical guidelines.
3. Clinical diagnosis of any mental health condition.
4. Current or former malignancy for which the participant has undergone resection, radiation therapy or chemotherapy within 5 years prior to baseline.
5. Diagnosis of any medical condition or disease, which in the opinion of the Principal Investigator (PI), may have either put the participant at risk, or influenced the results of the study or the participant's ability to participate in the study.
6. Diagnosis of any of the following medical conditions: HIV, COPD, severe/uncontrolled asthma, cystic fibrosis, bronchiectasis, interstitial lung disease, chronic renal failure, colon or small intestine problem, liver or kidney disease.
7. Currently enrolled or plan to be enrolled in another research study during the course of this investigation.
8. Planned or recent (within the last 12 months) bariatric surgery.
9. Current use of weight altering medication for the purpose of weight loss.
10. Uncorrected hypothyroidism or hyperthyroidism in the previous 12 months.
11. Alcohol or drug dependence during the previous 12 months.
12. Investigators and their immediate families. Immediate family was defined as a spouse, parent, child or sibling, whether biological or legally adopted.
13. Pregnant and/or breastfeeding.
14. Current smoker.
15. BMI ≥ 35.
16. Any other health risk that may have impaired the study's ability to assess the impact of nutrigenomic information to improve diet and health.

    -

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet quality | 8 weeks
  Healthy eating index

CONTACTS AND LOCATIONS:
Overall Officials: Karen Davison, PhD, Principal Investigator — Kwantlen Polytechnic University
Locations (1):
- Innovation Boulevard, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Araujo Almeida V, Littlejohn P, Cop I, Brown E, Afroze R, Davison KM. Comparison of Nutrigenomics Technology Interface Tools for Consumers and Health Professionals: A Sequential Explanatory Mixed Methods Investigation. J Med Internet Res. 2019 Jun 28;21(6):e12580. doi: 10.2196/12580. PMID 31254340
- [Derived] Littlejohn P, Cop I, Brown E, Afroze R, Davison KM. Comparison of Nutrigenomics Technology Interface Tools for Consumers and Health Professionals: Protocol for a Mixed-Methods Study. JMIR Res Protoc. 2018 Jun 11;7(6):e115. doi: 10.2196/resprot.9846. PMID 29891470